CLINICAL TRIAL: NCT05640765
Title: BeWell360-CG Care Model: Health and Wellness Coaching to Support Caregivers of Patients Living With Advanced Lung Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MC200201; NCI-2022-08655 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC200201 (Other: Mayo Clinic); 20-006003 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lung Carcinoma; Stage III Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods; Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: (Standard of care + Educational material) (Active Comparator): CGs receive the standard of care services assigned by the care team for their patient. Participants also receive additional educational and supportive material for health and wellness.
  Interventions: Other: Best Practice; Other: Educational Intervention; Other: Questionnaire Administration
- Arm 2: (Standard of care + BeWell360-CG) (Experimental): CGs receive the standard of care services assigned by the care team for their patient and participate in the BeWell360-CG coaching sessions on study.
  Interventions: Other: Best Practice; Other: Health Promotion and Education; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care services
  Other Names: standard of care; standard therapy
Other: Educational Intervention — Receive additional educational and supportive material
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm 1: (Standard of care + Educational material)
Other: Health Promotion and Education — Participate in BeWell360-CG Care Model sessions
  Arms: Arm 2: (Standard of care + BeWell360-CG)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial aims to develop a new care delivery model, called BeWell360-Care Giver (CG), to support caregivers of patients living with lung cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). The BeWell360-CG care model may enhance the wellbeing and quality of life of patients living with advanced lung cancer, and improve the current care standards for cancer patients and their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To pilot a novel, scalable, user-friendly health and wellness coaching (HWC) care model- the BeWell360-CG - that is embedded and integrated as part of a palliative approach to care for CGs of patients with advanced lung cancer.

II. To train palliative care (PC) staff to identify major themes and practical issues (barriers and facilitators) impacting CGs QoL and well-being, within and outside healthcare settings. (Aim 1) III. To evaluate the impact of BeWell360 on the CGs experience of their wellbeing and QoL. (Aim 2) IV. To evaluate the impact of BeWell360 on the quality of care of patients living with advanced lung cancer and receiving PC. (Aim 2) V. To create foundational knowledge about the feasibility and proof of concept of BeWell360-CG within PC for further future implementation and dissemination (translation) into practice. (Aim 3)

OUTLINE: Caregivers (CGs) are assigned to 1 of 2 arms.

ARM 1: CGs receive the standard of care services assigned by the care team for their patient. Participants also receive additional educational and supportive material for health and wellness.

ARM 2: CGs receive the standard of care services assigned by the care team for their patient and participate in the BeWell360-CG coaching sessions on study.

ELIGIBILITY:
Inclusion Criteria:

* CGs of patients with advanced lung cancer receiving care at Mayo Clinic Florida (MCF) in the Palliative Care (PC) or Oncology clinics
* Patient with a predicted life expectancy >=6 months
* Adult CGs' of any gender, race and ethnicity
* English speaking
* Willing to provide informed consent and complete HWC sessions, study interviews, and surveys. We will identify the respective patients through the patient appointment schedule list and use the patient electronic medical record (EMR) to confirm the point of contact of CGs.
* Palliative Care staff participating in the research study

Exclusion Criteria:

* Patients or CGs who are unable to complete surveys, coaching sessions and participate in interviews. Palliative Care clinicians will determine inability to participate based on burden to patient and clinical diagnosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Change in caregiver burden scores | 3-6 months
  Change in caregiver burden scores baseline, 3 months vs 6 months (or last follow-up) in caregivers as measured by burden-assessment scores [(e.g. Zarit Caregiver Burden, Palliative Score scale].

SECONDARY OUTCOMES:
Change in caregivers functional scores | Baseline to 6 months
  Change in caregivers functional scores (e.g. World Health Organization Disability Schedule [WHODAS]-12/36) from baseline versus (vs.) 6 months.
Change in caregivers' stress- and behavior-related scores | Baseline to 6 months
  Change in caregivers' stress- and behavior-related scores (e.g. Generalized Anxiety Disorder [GAD7]) from baseline vs. 6 months.
Change in Patient Health Questionnaire Depression (PHQ8) | Baseline to 6 months
  Change in caregivers' stress- and behavior-related scores (e.g. Patient Health Questionnaire Depression [PHQ8] from baseline vs. 6 months.
Change in patients Palliative Score (POS) | Baseline to 6 months
  Change in patients Palliative Score (POS) from baseline, 3 months vs. 6 months.
Change in patients Treatment burden (TBQ) scores | Baseline to 6 months
  Change in patients Treatment burden (TBQ) scores from baseline, 3 months vs. 6 months.
Perceptions of the BeWell360-Care Giver (CG) model | Baseline to 6 months
  Caregiver, patients, and clinicians' perceptions of the BeWell360-CG model using questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Moain Abu Dabrh, MB, BCh, Principal Investigator — Mayo Clinic; Maisha T. Robinson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials